CLINICAL TRIAL: NCT01072409
Title: Clinical Evaluation of the Nucleus 5 Cochlear Implant System
Brief Title: Clinical Evaluation of the Nucleus 5 Cochlear Implant (CI) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5255
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2014-09

CONDITIONS: Hearing Loss
Keywords: Speech perception ability in the CI alone condition
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): Single arm design
  Interventions: Device: Nucleus 5 Cochlear implant; Device: Cochlear implantation

INTERVENTIONS:
Device: Nucleus 5 Cochlear implant — Cochlear implant surgery
Device: Cochlear implantation — Implantation

SUMMARY:
To evaluate the performance of the Nucleus 5 Cochlear Implant System.

DETAILED DESCRIPTION:
Performance outcomes of newly implanted adult recipients using the Nucleus 5 Cochlear Implant System.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older at the time of the study.
* Postlinguistic onset of bilateral severe-to-profound sensorineural hearing loss
* Bilateral severe-to-profound hearing loss that meets current cochlear implant criteria (<50% open-set sentence recognition in quiet scores in the ear to be implanted and <60% in the best-aided condition)
* English spoken as the primary language.
* Willingness to participate in and to comply with all requirements of the study
* Subject may receive bilateral simultaneous cochlear implants.

Exclusion Criteria:

* Previous cochlear implant experience
* Congenital hearing loss (for the purpose of this study, onset prior to 2 years-of-age).
* Ossification, absence of cochlear development or any other cochlear anomaly that might prevent complete insertion of the electrode array.
* Normal hearing in one or both ears.
* Hearing loss of neural or central origin (e.g., deafness due to lesions on the acoustic nerve or central auditory pathway).
* Active middle-ear infection.
* Unwillingness and/or inability of the candidate to comply with all investigational requirements including, but not limited to, study protocol and surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Zwolan, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Implanted: Subjects who met study inclusion and completed the primary endpoint.
Period: Overall Study
Arm/Group | Implanted
Started | 45
Completed | 38
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Implanted
Number analyzed (Participants) | 38
Age, Continuous [Mean (Full Range); unit: years] | 63.6 [18 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20
Age at onset of hearing loss [Mean (Full Range); unit: years] | 40.8 [3 to 80]
Preoperative CNC word score - Treated ear [Mean (Standard Deviation); unit: percent correct] — The test consists of 10 lists with 50 monosyllabic words in each list. Subject responses are scored for both words and phonemes correct in the correct sequence. Subjects will be tested using a configuration of speech at 0º azimuth in quiet
  percent correct | 5.6 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: CNC Monosyllabic Word Performance - Treated Ear
Description: CNC Word Test is a validated test of open-set word recognition. The test consists of 10 lists with 50 monosyllabic words in each list. Subject responses are scored for both words and phonemes correct in the correct sequence. Subjects will be tested using a configuration of speech at 0º azimuth in quiet.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: percent correct
Arm/Group | Implanted
Number analyzed (Participants) | 38
percent correct | 56.8 (3.9)

ADVERSE EVENTS:
Arm/Group | Implanted
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No